CLINICAL TRIAL: NCT03083743
Title: A Randomized, Double-blind, Placebo-controlled in Parallel, Multicenter Phase III Trial of Recombinant Human Apo-2 Ligand for Injection（Dulanermin for Injection）in the Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: A Phase III Trial of Recombinant Human Apo-2 Ligand for Injection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Gebaide Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016L04304
Record Dates: First submitted 2017-02-28; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Non-small-cell Lung Cancer (NSCLC) Stage IV
Keywords: Carcinoma, Non-Small-Cell Lung; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Thoracic Neoplasms; Neoplasms; Lung Diseases; Antineoplastic Agents, Cytokines; Antineoplastic Agents; Biological activity factor; Genetic Engineering; Molecular Mechanisms of Pharmacological Action; Physiological Effects of Drugs
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Thoracic Neoplasms; Neoplasms; Lung Diseases | interventions — Injections; TNFSF10 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recombinant human Apo-2 ligand (Experimental): Recombinant human Apo-2 ligand for Injection
  Interventions: Biological: Recombinant human Apo-2 ligand for Injection
- Placebo (Placebo Comparator): Mimetic agent for recombinant human Apo-2 ligand for injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant human Apo-2 ligand for Injection — 150μg/kg/d IV (in the vein), on day 1 to 7 of each 21 day cycle
  Other Names: Dulanermin for injection
  Arms: Recombinant human Apo-2 ligand
Biological: Placebo — 150μg/kg/d IV (in the vein), on day 1 to 7 of each 21 day cycle
  Other Names: Mimetic for recombinant human Apo-2 ligand for injection
  Arms: Placebo

SUMMARY:
The trial is to evaluate the efficacy and safety of recombinant human Apo-2 ligand in treating patients with advanced retreated non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old
2. Pathologically diagnosed advanced non-small cell lung cancer (stage Ⅳ) with measurable lesions (diameter of tumor lesions displayed on CT scan ≥ 10 mm; short diameter of lymph node lesions on CT scan ≥ 15 mm; and no radiotherapy, radiofrequency ablation or other local treatment has been given to such measurable lesions)
3. Patients with negative EGFR or ALK gene-sensitive mutations or unknown status and with treatment failure or recurrence after previously undergoing the treatment with two chemotherapy regimens (at least one platinum-containing two-drug regimen included)
4. Patients with positive EGFR-TKI or ALK-TKI gene-sensitive mutations and with treatment failure or recurrence after previously undergoing one platinum-containing chemotherapy regimen may be included. Note that treatment given in neo-adjuvant therapy phase is not considered a part of the treatment regimen; however, if recurrence occurred within 6 months after the end of adjuvant therapy, the adjuvant therapy is considered a part of the treatment regimen, and if not within such 6 months, the adjuvant therapy is not considered a part of the treatment regimen.

   The term "treatment failure" is defined as: (1) progression presents in the course of treatment or after the last treatment with evidence of definitive imaging or clinical progression; (2) patients withdrawn from standard treatment due to inability to tolerate adverse events of grade IV and above hematological toxicity, of grade II and above non-hematological toxicity or of grade II and above major organ damage, such as heart, liver and kidney according to NCI-CTCAE Version 4.0.
5. ECOG status 0-1
6. Expected survival ≥ 3 months
7. Patients recovered from damages caused by other treatment given to them (≤ grade 1 according to NCI-CTCAE version 4.0); the interval of nitrosourea or mitomycin given was ≥ 6 weeks; the interval of other cytotoxic drugs, Avastin, radiotherapy or surgery was ≥ 4 weeks; and the interval of EGFR TKI molecular targeted drugs was ≥ 2 weeks
8. Major organs function normally, e.g. the following criteria are met (1) Blood routine tests shall comply with the criteria as follows (no transfusion of blood or blood products within 14 days, no correction with G-CSF and other hematopoietic stimulating factors):

   1. Hemoglobin（HB） ≥ 90 g/L
   2. Absolute neutrophil count（ANC） ≥ 1.5 × 10（9）/L
   3. Platelets（PLT ）≥ 80 × 10（9）/L

      (2) Biochemical test shall comply with the criteria as follows:

   <!-- -->

   1. Total bilirubin（TBIL） < 1.5 × upper limit of normal（ULN）
   2. Alanine aminotransferase （ALT） and aspartate aminotransferase（AST） <2.5 × ULN; and < 5 × ULN for patients with liver metastases
   3. Serum Cr ≤ 1.25 × ULN or endogenous creatinine clearance > 45 ml / min (Cockcroft-Gault formula)
9. Female patients at a childbearing age must have taken reliable contraceptive measures or received pregnancy test (either by serum or urine) showing a negative result within 7 days before inclusion and are willing to take appropriate contraceptive measures during the trial and in the following 8 weeks after the last administration of the test drug. Male patients shall agree to take appropriate contraceptive measures or have undergone surgical sterilization during the trial and in the following 8 weeks after the last administration of the test drug
10. Subjects shall participate in the study out of their own will, sign the informed consent, have good compliance, and cooperate with follow-up

    -

Exclusion Criteria:

1. Small cell lung cancer (including small cell carcinoma and mixed non-small cell lung cancer)
2. Patients who have a definitive history of severe allergy to biological products
3. Patients with active (without medical control) brain metastases, cancer meningitis, spinal cord compression, or with brain or leptomeninges disorders identified in CT or MRI examination in the inclusion process (however, patients with brain metastases who have completed treatment 21 days prior to the randomization and maintained symptomatic stability may be included)
4. Patients with Grade II and above myocardial ischemia or myocardial infarction and poorly controlled arrhythmia (including male patients with QTc interval ≥ 450 ms and female patients with QTc interval ≥ 470 ms)
5. Patients with Grade III to IV heart dysfunction according to NYHA or left ventricular ejection fraction (LVEF) <50% identified in cardiac ultrasound examination
6. Patients with persistent bradycardia and positive results in the atropine test
7. Patients with diseases concerning hemorrhagic tendency
8. Dropsy of serous cavity (including pleural effusion, ascites, and pericardial effusion) presenting clinical symptoms and requiring medical treatment
9. Patients with active hepatitis B or hepatitis C
10. Patients with active infection requiring anti-microbial treatment (such as antibiotics, antiviral drugs, and antifungal drugs)
11. Patients with a history of psychotropic drug abuse and failure to get rid of those drugs or who have mental disorders
12. Patients who have participated in other clinical trials regarding anti-tumor drugs within 4 weeks prior to randomization
13. Long-term users of adrenal cortex hormones or immunosuppressive agents
14. Patients with a history of or suffering from other non-cured malignancies, except for cured skin basal cell carcinoma, cervical carcinoma in situ and superficial bladder cancer
15. Pregnant or breastfeeding women; fertile patients who are unwilling or unable to take effective contraceptive measures
16. Patients with positive skin test results for injection of recombinant human Apo-2 ligand
17. Other conditions as the researcher consider that may have impacts on the performance of the clinical trial and interpretation of results

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival（OS） | From the date of randomization until the date of death from any cause, Assessed up to 36 months
  Survival information may be obtained via telephone contact with the patient, patients family or by checking the patients notes, hospital records, contacting the patients general practitioner or public death registry, where it is possible to do so under applicable local laws.

SECONDARY OUTCOMES:
Progression - free survival（PFS） | From date of randomization until the date of first documented progression or the date of death from any cause, whichever came first, evaluate once every six weeks (± 7 days) and assessed up to 36 months
  Progression Free Survival (PFS) : the time from start of study treatment to the first documentation of objective disease progression (PD) or death from any cause.
Objective Response Rate (ORR) | Every 6 weeks (± 7 days) up to 36 months
  Objective response rate: the percentage of subjects who have at least one visit response of CR or PR prior to any evidence of progression
Disease Control Rate (DCR) | Every 6 weeks (± 7 days) up to 36 months
  Disease control rate: the percentage of subjects who have at least one visit response of CR or PR or SD prior to any evidence of progression.
Quality of Life (QoL) | An evaluation is made every 3 weeks and until 30 days after the last medication

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Ph.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital，Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- See also: world cancer report 2014.WHO Keyword：Non-small Cell Lung Cancer — http://apps.who.int/bookorders/anglais/detart1.jsp?codlan=1&codcol=76&codcch=31
- See also: Journal title：Diagnosis and treatment of primary lung cancer (2011 edition)；2012/12 — http://www.cnki.net/